CLINICAL TRIAL: NCT04280419
Title: An Investigation of the Effect of Environmental Factors on Respiratory Muscle Endurance Test Results in Healthy Individuals
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Caner Acartürk, Physiotherapist, Hacettepe University
Other Study IDs: GO 19/71
Record Dates: First submitted 2019-05-29; First posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Healthy
Keywords: Motivational Music; respiratory muscle endurance; perceived exertion

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healty Subjects: Healthy Subjects Twenty-five healthy individuals will be included in the study. Physical properties of cases will be recorded. Respiratory functions and respiratory muscle strength will be evaluated. Physical activity will be assessed using the International Physical Activity Survey (IPAQ). Respiratory muscle endurance will be evaluated using an incremental workload test and fixed threshold load test. Tests will be repeated three times as motivational music, slow-paced music, and music. Heart rate, respiratory frequency, perceived exertion will be evaluated before and after the test.

SUMMARY:
This study aims to investigate the effect of music as an environmental factor on respiratory muscle endurance in healthy individuals.

DETAILED DESCRIPTION:
Respiratory muscles are as vital as the heart and can be susceptible to fatigue under certain conditions. Therefore, evaluation of the performance of respiratory muscles is critical in the event of impaired respiratory function. Respiratory muscle strength and respiratory muscle endurance tests are used for the evaluation of respiratory muscle functions. While measuring respiratory muscle strength provides information about the individual's pulmonary status, it cannot measure respiratory muscle strength. Respiratory muscle strength is the capacity of respiratory muscles to maintain a specific workload over time and is directly related to respiratory muscle fatigue.

Endurance of respiratory muscles can be evaluated by different methods such as sustained maximal ventilation, increased threshold load test, and fixed threshold load test, and there is no consensus on the best test.

Respiratory muscle fatigue in healthy individuals is known to complicate exercise performance. Fatigue of the respiratory muscles causes the accumulation of metabolites such as lactic acid in the muscles. In this case, the inspiratory respiratory muscle is activated in metaboreflexia; The firing frequency of afferent nerve fibers (type III and IV) increases. An increase in sympathetic stimulation causes general vasoconstriction. Exercise performance is adversely affected. This results in earlier termination of the exercise compared to the conditions where respiratory muscle fatigue is prevented. Therefore, it is stated that reducing or delaying metaboreflex may be an essential mechanism to improve exercise performance.

During general endurance exercise tests, it may be possible to change the environmental aspects (auditory stimuli, listen to motivational music, adjust the tempo with the metronome, give visual feedback, etc.) to suppress metaboreflexia and delay fatigue. It has been shown that listening to music during exercise reduces fatigue and reduces the perception of exercise in healthy individuals.

A possible explanation underlying the beneficial effects of sensory stimuli during exercise involves the integration of multiple physiological systems. In such cases, the attention and emotional effects of sensory stimuli can spread throughout the body by modulating pulmonary, cardiac, hormonal, and muscle systems. Although there are studies about the effects of music on healthy people during whole-body endurance exercises, the effect of music on respiratory muscle endurance was not investigated.

Therefore, this study aims to investigate the effect of music on respiratory muscle endurance test results.

ELIGIBILITY:
Inclusion Criteria:

1. Being 18-35 years old.
2. Volunteer to participate in the study.
3. Without any health problems.
4. To be cooperative with the tests to be done.

Exclusion Criteria:

1. To have an orthopedic, neurological, chronic cardiovascular, pulmonary, and systemic disease to prevent the tests from being performed.
2. To have a visual, auditory, or cognitive problem.
3. Not willing to participate in the study.
4. To have previous experience in music and instruments used in the study.
5. In the last three months, there is no history of exercise training.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Subjects
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-02-28 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscle endurance test | 1st 2 days
  Primary Outcome Measure:
  1.Respiratory muscle endurance test In our study, the muscle endurance test at the fixed threshold load with 24-hour intervals, and the muscle endurance test at the increased threshold load will be performed. Test times will be calculated and calculated in seconds. The result values will be obtained by multiplying the test time and the pressure value corresponding to the time. In the fixed threshold load, the respiratory muscle endurance test will be performed in 60% of the MIP. For testing, the nose will be closed with a clip after the device is placed in the mouth. The respiratory muscle endurance test will be started with 20% of the MIP in the increased threshold load. The pressure will be increased to 40%, 60%, 80%, and 100% respectively in two minutes intervals. The pressure change and the measurements made in this order shall be made without removing the device from the mouth. For testing, the nose will be closed with a clip after the device is placed.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No